CLINICAL TRIAL: NCT04388748
Title: Randomized Controlled Trial of Stress Management and Resiliency Training for Depression (SMART-D) vs Treatment as Usual in the Treatment of Major Depression
Brief Title: Stress Management and Resiliency Training for Depression vs Treatment as Usual in the Treatment of Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ashok Seshadri, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-009475
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMART-D Intervention Group (Experimental): Subjects will participate in Stress Management and Resiliency Training for Depression (SMART-D) therapy as well as treatment as usual which consists of any ongoing medication or psychotherapy based treatments that are currently in place.
  Interventions: Behavioral: Stress Management and Resiliency Training for Depression (SMART-D) Therapy
- Standard of Care Group (No Intervention): Treatment as usual will consist of any ongoing medication or psychotherapy based treatments that are currently in place.

INTERVENTIONS:
Behavioral: Stress Management and Resiliency Training for Depression (SMART-D) Therapy — 6 SMART-D group therapy sessions over 8 weeks
  Arms: SMART-D Intervention Group

SUMMARY:
Researchers are trying to find out if a Stress Management and Resiliency Training (SMART-D) therapy will help with major depression treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be enrolled for this study from patients attending the Mayo Clinic Depression Center, Mayo Clinic Family Medicine clinics, Behavioral Health and Primary Care Clinic at Mayo Clinic Health System, Austin, MN, with a diagnosis of major depression, in partial or near remission with PHQ-9 scores ≤14
* Participants will be required to be between 25 and 80 years old
* Able to speak English
* Able to provide written informed consent to participate in the study
* Participants must have DSM-V diagnostic confirmation of major depressive disorder (MDD) (American Psychiatric Association 2013).
* Participants will continue taking any prescribed medications from their clinical treatment team.
* Participants with co-morbid secondary diagnoses of persistent depressive disorder and generalized anxiety disorders will be included in the study.
* Participants must consent to audio recording of random group sessions which will be disclosed at the final study session.

Exclusion Criteria:

* Participants with bipolar disorder, active psychosis, active suicidal ideations, and active substance abuse meeting criteria for substance use disorders except nicotine, obsessive compulsive disorder, active panic disorder with agoraphobia or other phobic disorder, active posttraumatic stress disorder, active severe personality disorders will be excluded.
* Pregnant women - because of time duration of the study.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Change in patient health questionnaire depression assessment | Baseline, week 1, week 8, 3 months, 6 months
  Measured using the patient health questionnaire (PHQ-9) where total scores are reported on a scale of 1-4 Minimal depression, 5-9 Mild depression, 10-14 Moderate depression, 15-19 Moderately severe depression, 20-27 Severe depression
Change in severity of depression | Baseline, week 1, week 8, 3 months, 6 months
  Measured using the 17 item Hamilton Depression Rating scale (HAM-D) where total scores are reported on a scale of 0 - 7 = Normal, 8 - 13 = Mild Depression, 14-18 = Moderate Depression, 19 - 22 = Severe Depression, > 23 = Very Severe Depression

SECONDARY OUTCOMES:
Change in measures of resilience | 1 week, 8 week, 3 month, 6 month
  Measured using the Connor Davidson Resiliency Scale. Subjects are asked to indicate if they agree with 25 statements on a scale of 0=not true at all, 1=rarely true, 2=sometimes true, 3=often true and 4=true nearly all the time
Changed in perceived stress scale | 1 week, 8 week, 3 month, 6 month
  Measured using Perceived Stress Scale (PSS). Subjects are asked to answer a 10 question about their feelings and thoughts during the last month using a scale of 0 = Never, 1 = Almost Never, 2 = Sometimes, 3 = Fairly Often, 4 = Very Often

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Seshadri, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health System in Austin, Austin, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seshadri A, Fuller-Tyszkiewicz M, Harper L, Clark MM, Singh B, Chesak S, Kaur AS, McGillivray J, Frye MA. Randomized controlled trial of stress management and resiliency training for depression (SMART-D)-pilot study. PLoS One. 2025 Aug 19;20(8):e0328539. doi: 10.1371/journal.pone.0328539. eCollection 2025. PMID 40828809
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials